CLINICAL TRIAL: NCT03852745
Title: Managing Stress With Inflammatory Bowel Disease - an Open Trial of a Web-based Intervention
Brief Title: Managing Stress With Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2018:333; H2017:228 (Other: University of Manitoba)
Record Dates: First submitted 2018-08-01; First posted 2019-02-25 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2020-11

CONDITIONS: Inflammatory Bowel Disease; Anxiety; Depression
Keywords: cognitive behavioral therapy, online intervention
MeSH Terms: conditions — Inflammatory Bowel Diseases; Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: cognitive behavior therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy (Other): Online cognitive behavioral therapy intervention for 2 hours a week for 12 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — cognitive behavioral therapy; focus on learning skills including acceptance and commitment

SUMMARY:
This study will recruit persons with Inflammatory Bowel Disease. The investigators will contact people in an ongoing study (called IMAGINE) to recruit persons with high levels of stress, anxiety, or depression who are interested in a web-based program focused on skills in managing stress, anxiety and depression (a self-directed psychosocial intervention). The goal is to develop an internet-based psychosocial intervention to help persons with inflammatory bowel disease to cope with high levels of stress, anxiety or depression.

DETAILED DESCRIPTION:
Depression and anxiety are highly prevalent in IBD, with depression rates almost twice as high for those with IBD compared to the general community, and an estimated 30% overall with depression or anxiety. Perceived stress is a factor in the development of anxiety and depression. These comorbid conditions complicate management of IBD, adversely impacting patient outcomes and health, and increasing the resource burden to the health care system. However, comorbid depression and anxiety in IBD patients is undertreated, paralleling unmet mental health treatment needs in the general Canadian population. Development of alternate modes of effective treatment delivery is vital to enhance access, given limited mental health service availability. CBT has strong clinical evidence for its effectiveness in treating episodes of depression and anxiety as well as in preventing relapses. CBT may be successfully delivered as an internet-based intervention. While there are limited data on the efficacy of CBT tailored to the IBD population, studies targeting comorbid depression in IBD have resulted in significant mental health improvement. A recent study described an internet-based CBT for IBD reported modest outcomes (150), but participants were not selected to have psychiatric comorbidity and the primary outcomes were not improvement in mood or anxiety symptoms. The internet-based program used in this study will involve brief modules focused on areas important in managing stress, anxiety and depression including:

Core Topics: 1. About the Program, 2. IBD and Stress 3. Commitment to Living Life Fully, 4. The Brain-Gut Connection, 5. Understanding Anxiety, 6. Overcoming Avoidance, 7. Depression, 8. Behavioural Activation; Optional Topics: 9. Treatment Options, 10. IBD and the Workplace 11. Mindfulness

Procedures: Participants will be recruited with the use of a resources informing possible participants about the project. Patients expressing an interest in the program will receive a copy of the consent form for the study by email but asked not to sign it. They will be asked to schedule a time with the study coordinator to review with consent form, discuss any questions about the consent form or the program, and at the end to indicate verbally whether or not they provide consent. Those who provide consent will complete a brief psychiatric interview with the study coordinator to check for inclusion and exclusion criteria. The interview used will be the Mini International Neuropsychiatric Interview (MINI) for DSM5. Those who meet the inclusion criteria for the study will be sent a survey link to complete a the baseline measures for the program.Once participants are accepted into the study assessments will be completed at baseline, week 6, week 12, and during follow up at week 24.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with inflammatory bowel disease - Crohn's disease or ulcerative colitis
* A score on a scale measuring perceived stress, anxiety or depression indicating the presence of a clinically significant problem
* Regular access to a personal computer and Internet to allow access to the program
* Ability to read and write English

Exclusion Criteria:

* Presence of significant suicidal ideation or suicidal intent within the last six months
* Presence of self-harming behavior in the last six months
* Currently active substance use disorder (last six months)
* Psychotic disorder (last six months)
* Eating disorder (last six months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-18 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline, 6 weeks, 12 weeks, 24 weeks
  scale measuring anxiety and depression (14 items); likert scale 0 (not at all) to 3 (most of the time); higher scores(summed) indicate presence of anxiety or depression
Change in Perceived Stress Scale 4 (PSS-4) | Baseline, 6 weeks, 12 weeks, 24 weeks
  scale measuring psychological stress (4 items); likert scale 0 (never) to 4 (very often); higher scores indicate higher levels of perceived stress

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System - 29 (PROMIS-29) | Baseline, 6 weeks, 12 weeks, 24 weeks
  scale measuring health-related quality of life (29 items); likert scale 1 to 5, varying anchor points; in symptom oriented domains higher scores represent worse symptomology and in function oriented domains higher scores represent better functioning
Change in Clinical Global Impression - Improvement scale (CGI-I) | Baseline, 6 weeks, 12 weeks, 24 weeks
  scale measuring confidence in ability to manage stress (2 items); likert scale with varying anchor points; higher scores indicate higher stress and lower confidence
Change in the Work and Social Adjustment Scale (WSAS) | Baseline, 6 weeks, 12 weeks, 24 weeks
  scale measuring how inflammatory bowel disease impact daily functioning; likert scale 1(not at all) to 5 (very severely); higher scores indicate higher levels higher functional impairment
Change in Inflammatory Bowel Disease Symptom Inventory - Short Form (IBDSI) | Baseline, 6 weeks, 12 weeks, 24 weeks
  scale measuring symptoms of inflammatory bowel disease; likert scale with varying anchor points

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Furer, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba - College of Medicine, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No